CLINICAL TRIAL: NCT04165811
Title: Effects of Aerobic Dance Based Exercise Program on Lower Extremity Functions After Surgery in Obeses Awating Bariatric Surgery
Brief Title: Effects of Aerobic Dance Based Exercise Program After Surgery in Obeses Awating Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulfidan Tokgoz, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulU-C
Record Dates: First submitted 2019-11-14; First posted 2019-11-18 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2020-08

CONDITIONS: Morbid Obesity; Bariatric Surgery Candidate; Exercise; Obesity
Keywords: bariatric surgey; morbid obesity; aerobic exercise; lower extremity functions
MeSH Terms: conditions — Obesity, Morbid; Motor Activity; Obesity | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Dance based Exercise (Experimental): The exercise program will be administered 60 minutes, 2 days a week for 8 weeks. The exercise program will be created by physiotherapists as a group exercise program.
  Interventions: Other: Exercise treatment
- Counseling of physical activity (Experimental): Physical activity counseling is aimed at increasing the physical activity levels of the individuals who are waiting for bariatric surgery in the preoperative period.
  Interventions: Other: Counselling

INTERVENTIONS:
Other: Exercise treatment — A program consisting of aerobic dance based exercises and physical activity counseling accompanied by physiotherapists will be applied to the study group.
  Other Names: Aerobic dance based exercise
  Arms: Aerobic Dance based Exercise
Other: Counselling — Only physical activity counseling will be given to the subjects in this group.
  Other Names: Counseling of physical activity
  Arms: Counseling of physical activity

SUMMARY:
In this study, our primary aim is; investigate the effect of aerobic dance based exercise program on lower extremity functions (walking, stair stroke climbing, etc.) in obese individuals awaiting bariatric surgery.

DETAILED DESCRIPTION:
In this study, our primary aim is; investigate the effect of aerobic dance based exercise program on lower extremity functions (walking, stair stroke climbing, etc.) in obese individuals awaiting bariatric surgery. . Our secondary aim is to provide the individual with exercise habits and increase the level of physical activity in daily life with the exercise program planned according to the needs of the individual.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18-65
* Body mass index ≥40 or ≥35 with concomitant diseases
* No surgical operation in the last 6 months

Exclusion Criteria:

* Musculoskeletal disorders or systemic diseases that may prevent exercise
* The presence of psychiatric or neurological disease affecting cooperation and cognitive functions
* Presence of acute pain
* Heart pain
* Presence of previous myocardial infarction, subjective heart failure, uncontrolled diabetes and hypertension
* Regular exercise for 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-30 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Six Minute Walk Test | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  The Six Minute Walk Test was conducted according to a standardized protocol, using an internal hallway with the 30-meter distance marked by colored tape on the floor. Participants will be told that "the purpose of this test is to see how far you can walk in six minutes." Then, they will be instructed to "walk from end to end of the hallway at your own pace, in order to cover as much ground as possible." Participants will be allowed to stop and rest during the test, but will be instructed to resume walking as soon as they were able to do so. Before the walk started and at the end of the 6-min walk, participants will be shown a modified Borg dyspnea scale printed on a card and asked to "indicate your current degree of shortness of breath" on a scale of "0 = nothing at all" to "10 = very, very severe." At the end of the walk, they will be asked if they had experienced any of the following specific symptoms: dyspnea, chest pain, light-headedness, or leg pain, or any other symptoms.
Biodex Isokinetic Muscle Strength Measurement | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  sokinetic device. In all cases; In accordance with the test measurement protocol, both the Quadriceps Femoris and the Hamstring muscle strength were concentric contraction, primarily 5 repetitions at 60 ° / sec; then 10 repetitions at a rate of 240° / sec. After each limb measurement, a rest interval of 2 minutes will be given. Peak torque will be recorded in Newtonmeters / kilograms (Nm / kg)

SECONDARY OUTCOMES:
Bioelectrical Impedance Analysis-obesity score | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  Body components such as body fat percentage, body fat amount, lean body percentage, lean body mass, body water percentage, body water quantity, body mass index are calculated with bioelectrical impedance analysis. The muscle, fat and water ratio of the cases will be evaluated with Tanita Bioelectric Impedance Device. When the device assess the body fat percentage, body fat amount, lean body percentage, lean body mass, body water percentage, body water quantity and body mass index, it offers to us a score as called obesity score.
Biodex Balance System-Fall Risk Test | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  Biodex Balance System is a system that offers the possibility of evaluating the balance statically and dynamically. It is a system that measures the displacements in the center of gravity of a patient standing on an outpatient balance platform and the reactions of the support surface when the surface changes. For the static balance will be assessed with "Fall Risk Test " by using Biodex Balance system. Fall risk test offers to us a total score.
Evaluation of physical activity | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  The physical activity level of the cases will be evaluated with the International Physical Activity Questionnaire. In the questionnaire, the time spent by individuals in the last 7 days is questioned by considering the types of physical activity they perform in their daily lives. Met value of each activity is calculated to determine how active an individual is.
Sit and Up Test | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  The participant seated in a standard chair with a height of 43 cm with his arms crossed on his shoulders is asked to stand up and sit quickly for 30 seconds and the number of repetitions in which complete departure is achieved is recorded .
Stair Climbing Test | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  In the literature, it is seen that ladder up and down activity is evaluated by several different methods. One of the most commonly used methods is the ladder up and down test. The test person stops at the beginning of the ladder, after the order is given, the ladder starts to climb as fast as possible, and ends with the stopping of both feet at the beginning and the elapsed time is measured and recorded with a stopwatch. These measured values are used to evaluate the performance of a person going up and down stairs.
Impact of Weight on Quality of Life Questionnaire (IWQOL-Lite) | Change from baseline to 8 weeks follow up at two months and post-op 5 months
  The IWQOL (Weight Effect on Quality of Life Questionnaire) questionnaire is the first instrument intended to evaluate the quality of life specifically for obesity. It has been developed in the clinical setting for moderate to severe obesity and measures the quality of life aspects identified by obese people as the most important concerns in treatment. In the clinical evaluation of quality of life, when the necessity of short and obesity-specific tools is met, a more reduced form of the questionnaire, IWQOL-Lite, was developed.

CONTACTS AND LOCATIONS:
Overall Officials: Gülfidan Tokgöz, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No